CLINICAL TRIAL: NCT03541161
Title: Early Rehabilitation After Total Mastectomy and Immediate Reconstruction With Tissue Expander Insertion in Breast Cancer Patients
Brief Title: Early Rehabilitation After Immediate Reconstruction With TEI in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JiHye Hwang, Chairman, Physical & Rehabilitation Medicine Samsung Medical Center, Samsung Medical Center
Other Study IDs: SMC 2018-01-008-001
Record Dates: First submitted 2018-05-07; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Early rehabilitation; Conventional protocol; Tissue expander insertion
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early rehabilitation group: Breast cancer patients who underwent reconstructive surgery in samsung medical center from Jan 2017 to August 2017. Following early rehabilitation protocol, patients were educated to undergo a self-exercise program after short-term immobilization of 2 weeks.
- Conventional protocol group: Breast cancer patients who underwent reconstructive surgery in samsung medical center from May 2016 to Dec 2016. Following conventional protocol, patients were asked to immobilize their shoulder for more than 4 weeks and then undergo self-exercise program.

SUMMARY:
The purpose of the study is to find best post-operative rehabilitation protocol after total mastectomy and immediate reconstruction with tissue expander insertion. This study compared outcomes of two post-operative rehabilitation protocols ; "conventional protocol", which immobilized shoulder and upper arm motion for a month and "early rehabilitation protocol" with short-term immobilization period and early mobilization.

DETAILED DESCRIPTION:
To prevent surgical site complications, surgeons use so-called "conventional protocol", which immobilizes shoulder and upper arm motion for a month after total mastectmoy and immediate reconstruction with tissue expander insertion. To improve shoulder mobility and QOL of patients, the investigators introduced a new and early rehabilitation protocol with short-term immobilization in Jan 2017.

The investigators retrospectively reviewed total 115 breast cancer patients who underwent reconstructive surgery from May 2016 to Aug 2017. Patients who did their reconstruction before Jan 2017 followed conventional protocol and immobilized their shoulder for more than 4 weeks. Patients who did their reconstruction after Jan 2017 were educated to undergo a self-exercise program after short-term immobilization of 2 weeks. The investigators reviewed shoulder mobility, pain, QOL and complications at postoperative 1 month and 2 month in both group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has breast cancer
* Subject underwent total mastectomy and immediate reconstruction with tissue expander insertion

Exclusion Criteria:

* Patients who had pre-existing conditions before breast cancer surgery that limit shoulder movement.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients who underwent total mastectomy and immediate reconstruction with tissue expander insertion in samsung medical center by a plastic surgeon between May 2016 and August 2017
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The shoulder range of motion (ROM) | 2 month
  Shoulder ROM was measured in flexion, abduction, external rotation and internal rotation in the affected upper limb at post-operative 1 month and 2month. Measurements were conducted by a physiatrist using a goniometer with patients in seated position.
Surgical site complication | 2 month
  A plastic surgeon reviewed the surgical site for hematoma, seroma, surgical site infection, implant rupture, extrusion of the implant, asymmetry/displacement of the implant and any other complications at post-operative 1 month and 2month.

SECONDARY OUTCOMES:
Disabilities of arm, shoulder, and hand outcome measure questionnaire | 2 month
  The DASH questionnaire was used to assess shoulder function at postoperative 1 month and 2 month. Scores were transformed to a 0 to 100 scale.
Short-form 36 health survey | 2 month
  The SF36 was used to assess QOL at postoperative 1 month and 2 month. The SF36 contains 8 sections measuring 8 domains of QOL: physical functioning (PF), role limitations because of physical health problems (RP), bodily pain (BP), general health perception (GH), vitality (VT), social functioning (SF), role limitations because of emotional problems (RE), and mental health (MH). The 8 sections are summarized into a two-component summary: the physical component summary (PCS; PF, RP, BP, GH and VT) and mental component summary (MCS; MH, RE, SF, VT and GH).
Pain numeric rating scale | 2 month
  Self reported pain intensitiy at postoperative 1 month and 2 month. It scored 0-10 (0 = no pain; 10= pain as bad as can be)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hye Hwang, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim KH, Yeo SM, Cheong IY, Kim Y, Jeon BJ, Hwang JH. Early Rehabilitation after Total Mastectomy and Immediate Reconstruction with Tissue Expander Insertion in Breast Cancer Patients: A Retrospective Case-control Study. J Breast Cancer. 2019 Sep;22(3):472-483. doi: 10.4048/jbc.2019.22.e40. PMID 31598346

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03541161/Prot_SAP_000.pdf